EVALUATION OF SSS 1

## **Analysis Plan for:**

**Development and Pilot Trial of an Intervention to Reduce Disclosure Recipients Negative Social** 

**Reactions and Victims Psychological Distress and Problem Drinking** 

NCT03488927

Last approved August 25, 2020

**Contents:** 

**Analysis Plan** 

EVALUATION OF SSS 2

## **Analysis Plan**

Main effects. Treatment effect analyses compared participants in the intervention group who attended (Tx-Attender; n = 305) to both: (a) participants who were invited to the treatment but who did not attend (Tx-Nonattender; n = 531) and (b) participants in the control group (n = 432). We conducted ANCOVA analyses in SPSS. We added contrasts to compare the three groups using the /LMATRIX subcommand. Covariates included gender, year in college, and alcohol use in the past 30 days, based on baseline differences in these variables. We used these covariates for all models except those models including alcohol use frequency or binge drinking as moderators, where we only included gender and year in college (because there was no variability in alcohol use in the past 30 days with these moderators).

Dependent variables differed by hypothesis. To test Hypothesis 1, we compared the three groups on T2 intended reactions, among participants who responded about intentions at T2 (n = 415). To test Hypothesis 2, we compared the three groups on T2 actual reactions, among participants who responded about actual reactions at T2 (n = 474). To test Hypothesis 3, we compared the T2 scores on intermediary variables of all participants, with the T1 score of each outcome as a covariate to assess for differences in change.

Moderation analyses. We explored four categories of moderators: demographic, IPV/SA, alcohol use, and characteristics of actual disclosures. To explore moderation, intervention condition was operationalized via two dummy codes: Tx-Attender (1) vs. Control (0) and Tx-Attender (1) vs. Tx-Nonattender (0). We then entered these dummy-coded variables into a regression model in SPSS along with covariates consistent to the covariates in the main effect analysis, main effect of the moderator, and the two interactions of interest (i.e., interaction between each dummy-coded treatment variable and moderator). For example, for gender, we

EVALUATION OF SSS 3

included both gender  $\times$  Control and gender  $\times$  Tx-Nonattender in the model. Each moderator was tested separately. In cases of significant interactions, we used the SAS PROCESS macro to probe the direction of the interaction by looking at the simple effect of the intervention at both levels of dichotomous moderators and at high and low values ( $\pm$ 1 SD) of continuous moderators. We did not include moderators where the sample size of the group was five or fewer.